CLINICAL TRIAL: NCT00069459
Title: A 7 Month, Multicenter, Parallel, Double-Blind, Placebo-Controlled Comparison of 150-300 mg/Day of Extended-Release Bupropion Hydrochloride and Placebo for the Prevention of Seasonal Depressive Episodes in Subjects With a History of Seasonal Affective Disorder Followed by an 8-week Observational Follow-up Phase
Brief Title: Seasonal Affective Depression (SAD) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100006
Record Dates: First submitted 2003-09-25; First posted 2003-09-26 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Depressive Disorder
Keywords: Winter depression, winter blues, depression, seasonal depression, seasonal affective disorder
MeSH Terms: conditions — Depressive Disorder; Seasonal Affective Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Extended-release Bupropion Hydrochloride (Other): Extended-release Bupropion Hydrochloride
  Interventions: Drug: Extended-release Bupropion Hydrochloride

INTERVENTIONS:
Drug: Extended-release Bupropion Hydrochloride — Bupropion hydrochloride will be available in dose strength of 150 and 300 milligram (mg). Subjects will receive one tablet of 150 mg bupropion hydrochloride from Day 1 to 7, from Day 8 to Week 27 will receive one tablet of 300 mg bupropion hydrochloride and from Week 28-29 one tablet of bupropion hydrochloride

SUMMARY:
A placebo controlled study evaluating the effectiveness of medication in preventing winter depressive episodes in patients with a history of Seasonal Affective Disorder

DETAILED DESCRIPTION:
A 7-Month Multicenter, Parallel, Double-Blind, Placebo-Controlled Comparison of 150-300mg/day of Extended-release Bupropion Hydrochloride and Placebo for the Prevention of Seasonal Depressive Episodes in Subjects with a History of Seasonal Affective Disorder Followed by an 8-week Observational Follow-up Phase

ELIGIBILITY:
Inclusion Criteria:

* History of Major Depressive Disorder (MDD) with a seasonal pattern.

Exclusion Criteria:

* Current or past history of seizure disorder or brain injury.
* History or current diagnosis of anorexia nervosa or bulimia.
* Recurrent summer depression more frequently than winter depression.
* Primary diagnosis of panic disorder, Obsessive Compulsive Disorder (OCD), Post-traumatic Stress Disorder(PTSD), acute distress disorder, bipolar II disorder or other psychotic disorders.
* Initiated psychotherapy within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2003-09-23 (Actual); Primary Completion 2004-06-03 (Actual); Study Completion 2004-06-03 (Actual)

PRIMARY OUTCOMES:
End of season depression-free rate. | 7 months

SECONDARY OUTCOMES:
Time to onset of a seasonal depressive episode.Change from randomization on SIGH-SAD and HAMD-17. | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (44):
- United States (44):
  - GSK Investigational Site, Anchorage, Alaska
  - GSK Investigational Site, Hamden, Connecticut
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Wilmington, Delaware
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Edwardsville, Illinois
  - GSK Investigational Site, Hoffman Estates, Illinois
  - GSK Investigational Site, Northfield, Illinois
  - GSK Investigational Site, Oak Brook, Illinois
  - GSK Investigational Site, Oakbrook Terrace, Illinois
  - GSK Investigational Site, Cedar Rapids, Iowa
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Belmont, Massachusetts
  - GSK Investigational Site, Farmington Hills, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Kenilworth, New Jersey
  - GSK Investigational Site, Moorestown, New Jersey
  - GSK Investigational Site, Piscataway, New Jersey
  - GSK Investigational Site, Princeton, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Lawrence, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Lyndhurst, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Havertown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Lincoln, Rhode Island
  - GSK Investigational Site, Woodstock, Vermont
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Brown Deer, Wisconsin
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Menomonee Falls, Wisconsin
  - GSK Investigational Site, Middleton, Wisconsin

REFERENCES:
- [Result] Modell, JG, Rosenthal NE. Once-Daily Bupropion XL for the prevention of seasonal major depressive episodes. 43nd Annual Meeting of the American College of Neuropsychopharmacology, San Juan, Puerto Rico, 12-16 December, 2004.
- See also: Results for study 100006 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/100006?search=study&search_terms=100006#rs